CLINICAL TRIAL: NCT01423175
Title: Randomized, Multi-centre, Phase II Trial to Compare the Event-Free Survival of Clofarabine / Ara-C (ClAraC) or of FLAMSA Treatment in Patients With High Risk AML or Advanced MDS Scheduled for Allogeneic Stem Cell Transplantation
Brief Title: ClAraC or FLAMSA Followed by Stem Cell Transplantation to Treat High Risk AML or Advanced MDS
Acronym: ClAraC-SCT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hannover Medical School (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Principal Investigator, A. Ganser, Director of the Department of Hematology, Hemostasis, Oncology and Stem Cell Transplantation, Hannover Medical School
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ClAraC-SCT-01
Record Dates: First submitted 2011-08-24; First posted 2011-08-25 (Estimated); Last update posted 2011-08-29 (Estimated); Status verified 2011-08

CONDITIONS: Acute Myeloid Leukemia; MDS
Keywords: high risk acute myeloid leukemia; advanced myelodysplastic syndrome; allogenic stem cell transplantation; clofarabine
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Clofarabine; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ClAraC (Experimental)
  Interventions: Drug: Clofarabine, ara-C
- FLAMSA (Active Comparator)
  Interventions: Drug: FLAMSA

INTERVENTIONS:
Drug: Clofarabine, ara-C
  Arms: ClAraC
Drug: FLAMSA
  Arms: FLAMSA

SUMMARY:
ClAraC (consisting of one dose of clofarabine and ara-C for five days) or FLAMSA (consisting of one dose of fudarabine, amsacrine and ara-C for four days) will be administered followed by reduced-intensity conditioning regimen (RIC) in the setting of allogeneic stem cell transplantation (SCT). The aim of the study is to explore the antileukemic, immunosuppressive effects and toxicity and safety of clofarabine in combination with ara-C in the setting of RIC allogeneic transplantation compared with the FLAMSA-protocol for patients with high-risk acute myeloid leukemia (AML) or advanced myelodysplastic syndrome (MDS).

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent
2. Age > 18 at the day of inclusion
3. Patients with high risk AML or advanced MDS (IPSS score ≥ intermediate 2) scheduled for an allogeneic SCT from HLA-matched related or unrelated donor
4. Patients fulfilling at least one of the following risk factors:

   * Contraindication for conventional conditioning therapy
   * Relapsed or refractory to induction therapy
5. Adequate renal, hepatic and cardiac functions as indicated by the following values:

   * Serum creatinine ≤ 1.0 mg/dL; if serum creatinine > 1.0 mg/dL, then the estimated glomerular filtration rate (GFR) must be > 60 mL/min/1.73 m2
   * Serum bilirubin ≤ 1.5 x upper limit of normal (ULN)
   * Aspartate transaminase (AST) / alanine transaminase ALT) ≤ 2.5 x ULN
   * Alkaline phosphatase ≤ 2.5 x ULN
   * Left ventricular ejection fraction ≥ 50 %
6. Capable of understanding the investigational nature, potential risks and benefits of the study, and able to provide valid informed consent
7. Female patients of childbearing potential must have a negative serum pregnancy test at the day of inclusion
8. Female patients must meet one of the following criteria:

   * For female patients ≥ 50 years of age at the day of inclusion: Menopause since at least 1 year
   * Female patients < 50 years of age at the day of inclusion who meet all of the following criteria:

     * menopause since at least 1 year
     * serum FSH levels > 40 MIU/mL
     * serum estrogen levels < 30 pg/mL or negative estrogen test
   * 6 weeks after surgical sterilization by bilateral tubal ligation or bilateral ovariectomy with or without hysterectomy
   * Correct use of two reliable contraception methods from the time of screening and during the study for a minimum of 90 days after the last administration of study medication. This includes every combination of a hormonal contraceptive (such as oral, injection, transdermal patch, implant, cervical ring) or of an intrauterine device (IUD) with a barrier method (diaphragm, cervical cap, Lea contraceptive, femidom or condom) or with a spermicide. In case the patient takes hormone preparations for suppression of menstruation during the period of aplasia, a suitable and effective method of contraception has to be discussed with the investigator and used by the patient
   * General sexual abstinence from the time of screening, during the study until a minimum of 90 days after the last administration of study medication
   * Having only female sexual partners
   * Monogamous relationship with sterile male partner
9. Male patients must meet one of the following criteria:

   * 6 weeks after surgical sterilization by vasectomy
   * Correct use of two reliable contraception methods from the time of screening and during the study for a minimum of 90 days after the last administration of study medication. This includes every combination of a hormonal contraceptive (such as oral, injection, transdermal patch, implant, cervical ring) or of an intrauterine device (IUD) with a barrier method (diaphragm, cervical cap, Lea contraceptive, femidom or condom) or with a spermicide.
   * General sexual abstinence from the time of screening, during the study until a minimum of 90 days after the last administration of study medication
   * Having only male sexual partners
   * Monogamous relationship with sterile female partner

Exclusion Criteria:

1. Patients with acute promyelocytic leukemia with t(15;17)
2. Current concomitant chemotherapy, radiation therapy, or immunotherapy other than as specified in the protocol
3. Any anticancer therapy within 2 weeks before study entry with the exception of hydroxyurea. The patient must have recovered from all acute toxicities from any previous therapy
4. Current participation in any other clinical trial and/or participation in another clinical trial within 30 days before the trial begins
5. Have any other severe concurrent disease, or have a history of serious organ dysfunction or disease involving the heart (heart insufficiency ≥ NYHA II), kidney (serum creatinine > 1.5 x normal serum level), liver (bilirubin > 1.5 x normal serum level, AST / ALT, AP > 2.5 x normal serum level), or other organ system that may place the patient at undue risk to undergo treatment
6. Patients with a systemic fungal, bacterial, viral, or other infection not controlled (defined as exhibiting ongoing signs/symptoms related to the infection and without improvement, despite appropriate antibiotics or other treatment)
7. Human immunodeficiency virus (HIV) positivity
8. Pregnant or lactating patients
9. Any significant concurrent disease, illness, or psychiatric disorder that would compromise patient safety or compliance, interfere with consent, study participation, follow up, or interpretation of study results
10. Have had a diagnosis of another malignancy, unless the patient has been disease-free for at least 3 years following the completion of curative intent therapy, with the following exceptions:

    * Patients with treated non-melanoma skin cancer, in situ carcinoma, or cervical intraepithelial neoplasia, regardless of the disease-free duration, are eligible for this study if definitive treatment for the condition has been completed
    * Patients with organ-confined prostate cancer with no evidence of recurrent or progressive disease based on prostate-specific antigen (PSA) values are also eligible for this study if hormonal therapy has been initiated or a radical prostatectomy has been performed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-07; Primary Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
Event-free survival

SECONDARY OUTCOMES:
Overall survival
Morbidity after allogeneic SCT with focus on cardiac toxicity
Rate of engraftment
Kinetics of chimerism after allogeneic SCT
Relapse-free survival
Mortality after allogeneic SCT with focus on cardiac toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Arnold Ganser, Prof. Dr., Principal Investigator — Hannover Medical School
Locations (3):
- Germany (3):
  - Hannover Medical School, Hanover
  - Universitaetsklinikum des Saarlandes, Homburg/Saar
  - Universitaetsklinikum Leipzig AoeR, Leipzig